CLINICAL TRIAL: NCT01048086
Title: 90Y-DOTA-tyr3-Octreotide With or Without Retinoic Acid for the Treatment of Neuroblastoma and Neuroendocrine Tumors in Children and Young Adults. A Randomized, Placebo Controlled Phase II Trial With Dosimetry Guided Dosing
Brief Title: 90Y DOTA/Retinoic Acid for Neuroblastoma and Neuroendocrine Tumor (NET)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were enrolled because the company that pledged the drug does not yet have it available.
Sponsor: University of Iowa (Other)
Collaborators: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, O'Dorisio, M S, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200904707
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Neuroblastoma; Neuroendocrine Tumor
Keywords: neuroblastoma; neuroendocrine tumor; NET; retinoic acid
MeSH Terms: conditions — Neuroblastoma; Neuroendocrine Tumors | interventions — Tretinoin; Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retinoic Acid (Experimental)
  Interventions: Drug: Retinoic Acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retinoic Acid — 160 mg, given orally, divided BID on Days 1-4 of each cycle for 4 cycles. Each cycle will be six weeks in duration. Dose will be adjusted to 5.33 mg/kg/day divided BID for children <12 kg.
  Other Names: 13-cis retinoic acid
  Arms: Retinoic Acid
Drug: Placebo — Placebo will be given in the same manner as retinoic acid in capsules that look identical.
  Arms: Placebo

SUMMARY:
This study is for patients with neuroblastoma or a neuroendocrine tumor who have not been able to have standard therapy or have failed the first-line therapy. The purpose of this study is to assess the safety and effectiveness of the combination of retinoic acid and Onalta (Y-90-DOTA-tyr3-Octreotide) in treating neuroblastoma and neuroendocrine tumors.

DETAILED DESCRIPTION:
This study builds on the promising results of the Phase I trial of 90Y-DOTA-tyr3-Octreotide in childhood solid tumors and the history of cis-Retinoic Acid (cis-RA) use in children with neuroblastoma. This study will combine these two agents in a randomized Phase II trial. The safety and feasibility of using individual dosimetry measurements to maximize the 90Y-DOTA-tyr3-Octreotide radiation dose to tumor while limiting the renal radiation dose to 23 Gy will be rigorously tested.

Fixed dosing will allow each subject to receive three cycles of 90Y-DOTA-tyr3-Octreotide at 50 mCi/m2. Dosimetry will be performed at each of these cycles; the combined dosimetry measurements will be utilized to determine whether or not a fourth cycle will be administered and, if so, what that dose will be. The administration of this additional cycle is conditional upon a) a subject not experiencing a dose-limiting toxicity during any previous cycle and b) meeting all criteria required at study initiation prior to the fourth dose.

ELIGIBILITY:
Inclusion Criteria:

1. Disease Criteria

   1. A pathologically confirmed (histology or cytology) malignant neoplasm that is determined to be neuroblastoma or neuroendocrine tumor. The subject's neoplastic disease must have been (positively) imaged by OctreoScan® or 111In-DOTA-tyr3-Octreotide within 4 weeks prior to ordering study drug.
   2. b) Disease not amenable to standard treatment (disease present after surgery and/or Sandostatin treatment) or subject has failed existing first line therapy (surgery and chemotherapy/radiation therapy).
   3. c) Upon baseline disease assessment, all subjects must have at least 1 measurable, evaluable, site of disease that either has never been irradiated or has been previously irradiated and has since demonstrated progression based on COG response criteria. Children's Oncology Group response criteria include: 1) Complete response (CR) is defined as no measureable disease; 2) partial response (PR) as >50% decrease in longest X widest perpendicular diameter of target lesions with no increase in any lesions and no new lesions; 3) minor response (MR) as >25%<50% decrease in target lesions with no increase in any lesion and no new lesions; 4) stable disease as <25% increase or decrease in any target lesion and no new lesions; 5) Progressive disease (PD) as an increase >25% in any measureable lesion or the presence of any new lesion was considered progressive disease (PD). Response will be assessed based on intent to treat for all subjects who receive at least one dose of 90Y-DOTA-tyr3-Octreotide.
   4. Each subject must have at least one measurable somatostatin receptor positive lesion that has not had local irradiation via external beam, conformal or stereotactic radiation treatments within 4 weeks prior to study drug administration and no full craniospinal radiation within 3 months prior to study drug administration.
   5. Bone marrow with >/= 40% cellularity or with 1 million CD34+ stem cells/kg stored.
   6. Life expectancy > 2 months and < 12 months.
   7. Biopsy of at least one lesion or bone marrow that has been identified as progressive malignancy within four weeks prior to the first dose of Onalta® is encouraged but not required. If no biopsy can be performed for clinical reasons, available tissue from a previous biopsy will be required.
2. Age 6 months-30 years.
3. COG performance status /= 60% or Lansky Play Scale >/= 60%).
4. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count >1000/mm3
   * platelets >100,000/mm3
   * total bilirubin <1.5 x nl for age and weight
   * AST(SGOT) & ALT(SGPT) <2.5 X institutional upper limit of normal for age
   * creatinine <1.0 for children <5 years of age; <1.2 for children 5-10 years of age; <1.7 for >10 years AND
   * GFR >80 mL/min/1.73 m2
   * urinalysis with no greater than 1+ hematuria or proteinuria
5. Cardiac function must be adequate

   * shortening fraction of > 28% by echo
   * ejection fraction > 50% by bi-plane method of echo
6. The effects of 90Y-DOTA-tyr3-Octreotide on the developing human fetus are unknown. Retinoic acid is known to be harmful to the developing human fetus. For these reasons and because Class C agents are known to be teratogenic, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Serum triglycerides <300 mg/dL.
9. Concomitant Therapy - The subject may not receive any other approved or investigational anti-neoplastic therapies for the treatment of the refractory somatostatin-receptor positive tumor during the course of the study, excluding somatostatin analogues and bisphosphonates. However, all subjects on somatostatin analogue therapy will discontinue therapy from 12 hours prior to a) injection with OctreoScan® or 111In-DOTA-tyr3-Octreotide, and b) infusion with 90Y-DOTA-tyr3-Octreotide until 12 hours post administration. Subjects who have been on hormonal therapy (other than somatostatin analogues) for > 2 months with SD or PD may continue to receive hormonal therapy during this study. Subjects who initiate another tumor-specific therapy will be discontinued from further treatment with 90YDOTA-tyr3-Octreotide. Disease progression alone does not mandate discontinuation of a subject from treatment.

All subjects who have received at least one dose of 90Y-DOTA-tyr3-Octreotide must continue into the Long-Term Follow-up Study Period at the point of treatment discontinuation. This is necessary to determine any long-term effects of treatment with 90Y-DOTA-tyr3-Octreotide. Subjects may receive, at the discretion of the investigator, appropriate medical treatment for medical problems that arise while on study.

Exclusion Criteria for enrollment and Cycle One study period:

1. Age less than 6 months or greater than 30 years.
2. Pregnancy or breast feeding.
3. Surgery, radiation or chemotherapy within 4 weeks of study drug administration.
4. Another investigational drug within 4 weeks of study drug administration.
5. More than one, concurrent, malignant disease.
6. History of congestive heart failure, unless cardiac ejection fraction ≥ 40%.
7. Another significant medical, psychiatric, or surgical condition which is currently uncontrolled by treatment and which would likely affect the subject's ability to complete this protocol.
8. Any subject for whom, in the opinion of their physician, a 24-hour discontinuation of somatostatin analogue therapy represents a health risk. Also subjects who have received long-acting somatostatin analogue in the past 21 days are excluded.
9. Bone marrow cellularity <40% without >/= 1 million CD34+ stem cells/kg stored.
10. External beam radiation to both kidneys (scatter doses of < 500 cGy to a single kidney or radiation to < 50% of a single kidney is acceptable).
11. Antibodies to 90Y-DOTA-tyr3-Octreotide or Octreotide.
12. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of study drug administration or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
13. Patients may not be receiving any other investigational agents.
14. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 90YDOTA-tyr3-Octreotide.
15. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
16. Pregnant women are excluded from this study because 90Y-DOTA-tyr3-Octreotide is a Class C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 90Y-DOTA-tyr3-Octreotide, breastfeeding should be discontinued if the mother is treated with 90Y-DOTA-tyr3-Octreotide.
17. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with 90Y-DOTA-tyr3-Octreotide. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluate tumor response to 90Y-DOTA-tyr3-Octreotide alone and in combination with 13-cis retinoic acid for the treatment of children and young adults with recurrent, somatostatin-receptor positive tumors | 6 weeks after last treatment

SECONDARY OUTCOMES:
Estimate and compare time to tumor progression and overall survival in the patients treated with 90Y-DOTA-tyr3-Octreotide alone and in combination with 13-cis retinoic acid. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: M Sue O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States